CLINICAL TRIAL: NCT06918431
Title: A Phase 2 Study Evaluating the Safety and Efficacy of Asparaginase Erwinia Chrysanthemi- Recombinant-Rywn (Recombinant Erwinia Asparaginase) During Pediatric-Inspired Regimen in High-Risk Adults With Newly Diagnosed ALL or LBL
Brief Title: Asparaginase Erwinia Chrysanthemi With Chemotherapy for the Treatment of High-Risk Adults With Newly Diagnosed Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24442; NCI-2025-02184 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24442 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: B Acute Lymphoblastic Leukemia, Philadelphia Chromosome Negative; Lymphoblastic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — asparaginase erwinia chrysanthemi recombinant; Asparaginase; Specimen Handling; Biopsy; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Spinal Puncture; Mercaptopurine; azathiopurine; Methotrexate; merphos; Magnetic Resonance Spectroscopy; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (asparaginase Erwinia chrysanthemi) (Experimental): See Detailed Description
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Procedure: Echocardiography; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Positron Emission Tomography; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Asparaginase Erwinia chrysanthemi — Given IM
  Other Names: Asparaginase Erwinia chrysanthemi (Recombinant)-rywn; Asparaginase Erwinia chrysanthemi, Recombinant-rywn; Asparaginase Erwinia chrysanthemi-rywn; Crisantaspase; Crisantaspase Biobetter JZP-458; Crisantaspasum; Enrylaze; Erwinase; Erwinaze; JZP 458; JZP-458; JZP458; PF743; RC-P JZP-458; Recombinant Asparaginase erwinia chrysanthemi JZP-458; Recombinant Crisantaspase JZP-458; Recombinant Erwinia asparaginase JZP-458; Rylaze
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and/or biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and/or biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Cytarabine — Given IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Cytarabine — Given IV or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial tests the safety, side effects, and effectiveness of asparaginase Erwinia chrysanthemi during induction chemotherapy followed by consolidation chemotherapy in treating high-risk adults with newly diagnosed acute lymphoblastic leukemia or lymphoblastic lymphoma. Asparaginase Erwinia chrysanthemi, a type of protein synthesis inhibitor, is a drug that is made up of the enzyme asparaginase, which comes from the bacterium Erwinia chrysanthemi, and is used with other drugs in people who cannot take asparaginase that comes from the bacterium E. coli. Asparaginase Erwinia chrysanthemi breaks down the amino acid asparagine and may stop the growth of cancer cells that need asparagine to grow. It may also kill cancer cells. Induction therapy, consisting of cytarabine, dexamethasone, vincristine, daunorubicin, methotrexate, and rituximab, is the first choice of treatment. Consolidation therapy, consisting of cyclophosphamide, cytarabine, vincristine, mercaptopurine, methotrexate and rituximab, is given after initial therapy to kill any remaining cancer cells. Vincristine is in a class of medications called vinca alkaloids. It works by stopping cancer cells from growing and dividing and may kill them. Methotrexate is in a class of medications called antimetabolites. It is also a type of antifolate. Methotrexate stops cells from using folic acid to make deoxyribonucleic acid (DNA) and may kill cancer cells. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill cancer cells. It may also lower the body's immune response. Cytarabine and mercaptopurine stop cells from making DNA and may kill cancer cells. They are a type of antimetabolite. Daunorubicin blocks a certain enzyme needed for cell division and DNA repair and may kill cancer cells. It is a type of anthracycline antibiotic and a type of topoisomerase inhibitor. Dexamethasone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Giving asparaginase Erwinia chrysanthemi with induction chemotherapy followed by consolidation chemotherapy may be safe, tolerable, and/or effective in treating high-risk adults with newly diagnosed acute lymphoblastic leukemia or lymphoblastic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of asparaginase Erwinia chrysanthemi (asparaginase Erwinia chrysanthemi-recombinant-rywn [recombinant Erwinia asparaginase]; 25 mg/m^2 every 48 hours [hrs]) as first asparaginase during induction therapy through the assessment of type, frequency, severity, attribution, time course and duration of adverse events. (Safety Lead-in) II. To evaluate the proportion of patients with grade 3 or higher (G3+) hepatotoxicity that are at least possibly related to the study drug (recombinant Erwinia asparaginase) and not resolved to grade 1 or lower within 14 days of occurrence in the target patient population during induction. (Expansion)

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of recombinant Erwinia asparaginase (25 mg/m^2 every 48 hrs) as first asparaginase during induction therapy through the assessment of type, frequency, severity, attribution, and duration of adverse events (expansion cohort).

II. To evaluate composite complete remission (CR or CR with incomplete hematologic recovery [CRi]) rate after induction ± extended induction.

III. To evaluate CR rate after induction ± extended induction. IV. To evaluate minimal residual disease (MRD) negativity rate after induction ± extended induction.

V. To evaluate number of patients able to receive extended induction or post induction consolidation or salvage therapy within 42 days from initiating induction.

VI. To evaluate MRD negativity rate after consolidation for patients receiving the study drug.

VII. To evaluate the proportion of patients with G3+ hepatotoxicity that are at least possibly related to the study drug during induction.

VIII. To evaluate the proportion of patients maintaining adequate 48 hour nadir serum asparaginase activity (NSAA ≥ 0.1 IU/mL) post recombinant Erwinia asparaginase during induction +/- extended induction.

IX. To evaluate the duration of G3+ hepatotoxicity.

EXPLORATORY OBJECTIVES:

I. To evaluate the safety and tolerability of recombinant Erwinia asparaginase (at approved dosing) as first asparaginase during extended induction and consolidation therapy through the assessment of type, frequency, severity, attribution, time course and duration of adverse events.

II. To evaluate the proportion of patients maintaining adequate, either at 48 hours or 72 hrs, nadir serum asparaginase activity (NSAA ≥ 0.1 IU/mL) post recombinant Erwinia asparaginase during consolidation.

III. To evaluate the molecular profile by next-generation sequencing (NGS) and its association with MRD- response to recombinant Erwinia asparaginase based induction.

OUTLINE:

INDUCTION (CYCLE 1): Patients receive cytarabine intrathecally (IT) on day 1, dexamethasone orally (PO) twice daily (BID) on days 1-7 and 15-21, vincristine intravenously (IV) on days 1, 8, 15, and 22, daunorubicin IV over 5-30 minutes on days 1, 8, 15, and 22, asparaginase Erwinia chrysanthemi intramuscularly (IM) on days 4, 6, 8, 10, 12, 14, and 16, and methotrexate IT on days 8 and 29. Patients with CNS3 disease also receive methotrexate IT on days 15 and 22. CD20 positive patients also receive rituximab IV on day 8. Treatment continues for 4 weeks in the absence of disease progression or unacceptable toxicity. Patients with M2 marrow (> 5% lymphoblasts) on day 29 proceed to Extended Induction Cycle 1A. All other patients proceed to Consolidation Cycle 2.

EXTENDED INDUCTION (CYCLE 1A): Patients receive dexamethasone PO BID on days 1-7, vincristine IV on days 1 and 8, daunorubicin IV over 5-30 minutes on day 1, and asparaginase Erwinia chrysanthemi IM on days 4, 6, 8, 10, 12, 14, and 16 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION (CYCLE 2): Patients receive cyclophosphamide IV on days 1 and 29, cytarabine IV or subcutaneously (SC) on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO on days 1-14 and 29-42, vincristine IV on days 15, 22, 43, and 50, and methotrexate IT on days 1, 8, 15 and 22 (NOTE: Patients with CNS3 disease omit methotrexate on days 15 and 22). CD20 positive patients also receive rituximab IV on days 1 and 20. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit may also receive asparaginase Erwinia chrysanthemi IM every other day on days 15, 17, 19, 21, 23, 25, 27, 43, 45, 47, 49, 51, 53, and 55 or every Monday/Wednesday/Friday (if days 15 and 43 are Mondays) on days 15, 17, 19, 22, 24, 26, 43, 45, 47, 50, 52, and 54 at discretion of treating physician. Patients may receive 2 courses of every other day or Monday/Wednesday/Friday treatment in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo echocardiography at screening and blood sample collection, bone marrow aspiration and/or biopsy, lumbar puncture, and computed tomography (CT) and/or positron emission tomography (PET)/CT throughout the study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age between 18 and 39 with body mass index (BMI) ≥ 30 or age 40-54 years, regardless of BMI
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Patients with newly diagnosed Philadelphia (Ph)-negative (-) acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma (LBL) according to World Health Organization (WHO) criteria

  * Both B- and T-cell phenotypes are allowed.
* CD20+ patients only: White blood cell count less than 25 x 10^9/L prior to initiation of rituximab (within 14 days prior to day 1 of protocol therapy)

  * Cytoreduction with hydroxyurea or steroid or a single dose of intrathecal chemotherapy prior to treatment may be required
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (within 14 days prior to day 1 of protocol therapy) (unless has Gilbert's disease or related to underlying leukemia, ≤ 3 x ULN)
* Aspartate aminotransferase (AST) ≤ 3.0 x ULN (AST ≤ 5.0 x ULN if related to underlying leukemia) (within 14 days prior to day 1 of protocol therapy)

  * Note: AST ≤ 3.0 x ULN at the time of first dose of recombinant Erwinia asparaginase administration
* Alanine aminotransferase (ALT) ≤ 3.0 x ULN (ALT ≤ 5.0 x ULN if related to underlying leukemia) (within 14 days prior to day 1 of protocol therapy)

  * Note: ALT ≤ 3.0 x ULN at the time of first dose of recombinant Erwinia asparaginase administration
* Creatinine clearance of ≥ 60 mL/min per 24-hour urine test or the Cockcroft-Gault formula (within 14 days prior to day 1 of protocol therapy)
* Prothrombin (PT) ≤ 1.5 ULN (within 14 days prior to day 1 of protocol therapy)
* Activated partial thromboplastin time (aPTT) ≤ 1.5 ULN (within 14 days prior to day 1 of protocol therapy)
* Left ventricular ejection fraction (LVEF) ≥ 50%

  * Note: Echocardiogram to be performed within 42 days prior to day 1 of protocol therapy
* Seronegative for active hepatitis B virus (HBV) (surface antigen negative and anti-hepatitis B virus core antibody [HBc] negative) for CD20+ patients only

  * Note Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (within 14 days prior to day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective (non-hormonal) method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy. For participants taking rituximab, effective birth control or abstinence to be used for at least 12 months after last dose

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Leukemia-based therapy with chemotherapy with the exception of:

  * Cytoreduction with steroid or hydroxyurea or a single dose of intrathecal chemotherapy is allowed before initiating the study
  * Prior treatment with all-trans-retinoic acid (ATRA) for suspected acute promyelocytic leukemia (APL) is allowed
* Received previous treatment with any other asparaginase formulation
* Must not have received or planning to receive live vaccine while being on study or 2 weeks before and after completion of treatment. For CD20+ patients only: Must not have received any vaccines (live or non-live) 4 weeks before rituximab
* Known presence of Philadelphia chromosome positive (Ph+; t[9;22])
* Class III/IV cardiovascular disability according to the New York Heart Association classification. Subjects with controlled, asymptomatic atrial fibrillation can enroll
* Parenchymal central nervous system (CNS) involvement
* Participants with clinically significant arrhythmia or arrhythmias not stable on medical management within two weeks of enrollment
* History of acute cardiovascular ischemic event, i.e., myocardial infarction or unstable angina within 6 months of enrollment
* History of intracranial thrombosis or history of recurrent thrombosis or grade 3 and greater pulmonary embolism (except for catheter-related thrombosis)
* Participants with history of grade ≥ 3 pancreatitis
* History of alcohol overuse if deemed relevant in investigator opinion
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Uncontrolled active infection
* Clinically significant uncontrolled illness
* Other active malignancy
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) (Safety Lead-in) | Up to completion of induction cycle (cycle length = 28 days)
  Will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Will be summarized for evaluable patients in terms of type (organ affected or laboratory determination), severity, time of onset, duration, frequency, probable association with the study treatment and reversibility or outcome.
Incidence of unacceptable adverse events (Safety Lead-in) | Up to completion of induction cycle 1 (cycle length = 28 days)
  Will be summarized for evaluable patients in terms of type (organ affected or laboratory determination), severity, time of onset, duration, frequency, probable association with the study treatment and reversibility or outcome.
Incidence of grade 3 or higher hepatotoxicity and not resolved to grade 1 or lower within 14 days of occurrence (Expansion) | Up to completion of induction (cycle length = 28 days)
  Will be graded using NCI CTCAE v 5.0. Will be summarized for evaluable patients in terms of type (organ affected or laboratory determination), severity, time of onset, duration, frequency, probable association with the study treatment and reversibility or outcome. The overall rate and its 95% Clopper Pearson binomial confidence interval (CI) will be estimated.

SECONDARY OUTCOMES:
Incidence of AEs (Expansion cohort only) | Up to completion of induction (cycle length = 28 days)
  Will be graded according to NCI CTCAE v 5.0. Will be summarized for evaluable patients in terms of type (organ affected or laboratory determination), severity, time of onset, duration, frequency, probable association with the study treatment and reversibility or outcome.
Composite complete response (CR) | After induction with or without extended induction (induction cycle length = 28 days, extended induction cycle length = 16 days)
  Will be defined as CR and CR with incomplete hematologic recovery. The overall rate and its 95% Clopper Pearson binomial confidence interval (CI) will be estimated.
CR rate | After induction with or without extended induction (induction cycle length = 28 days, extended induction cycle length = 16 days)
  The overall rate and its 95% Clopper Pearson binomial confidence interval (CI) will be estimated.
Minimal residual disease (MRD) negativity | After induction with or without extended induction (induction cycle length = 28 days, extended induction cycle length = 16 days), at day 28 +/- 42
  Will be defined as residual leukemia < 0.01% by flow cytometry and/or clonoSEQ. The overall rate and its 95% Clopper Pearson binomial confidence interval (CI) will be estimated.
MRD negativity | After consolidation (consolidation cycle length = 8 weeks)
  The overall rate and its 95% Clopper Pearson binomial confidence interval (CI) will be estimated.
Proportion of patients to receive extended induction/consolidation/salvage therapy | Within 42 days from initiating induction
  The overall rate and its 95% Clopper Pearson binomial confidence interval (CI) will be estimated.
Incidence of grade 3 or higher hepatotoxicity | During induction (cycle length = 28 days)
  The overall rate and its 95% Clopper Pearson binomial confidence interval (CI) will be estimated.
Nadir serum asparaginase activity (NSAA) | At 48 hours post Erwinia asparaginase during induction +/- extended induction (induction cycle length = 28 days, extended induction cycle length = 16 days)
  Will be defined as NSAA >= 0.1 IU/mL. The overall rate and its 95% Clopper Pearson binomial confidence interval (CI) will be estimated.
Duration of grade 3 or higher hepatotoxicity | Time from starting date of the grade 3 or higher hepatoxicity to the resolving (grade ≤ 1) date, assessed up to 30 days after last dose of study treatment
  Will be summarized by descriptive statistics (mean, range, etc).

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Aldoss, Principal Investigator — City of Hope Medical Center
Locations (8):
- United States (8):
  - City of Hope at Phoenix, Phoenix, Arizona
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio